CLINICAL TRIAL: NCT05946096
Title: Effects of Dynamic Surface Exercise Training on Trunk Control and Gross Motor Functions in Children With Diplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ayesha Hameed (Other)
Responsible Party: Sponsor-Investigator, Ayesha Hameed, Researcher, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULahore123
Record Dates: First submitted 2023-04-09; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Cerebral Palsy Spastic Diplegia
Keywords: trunk control; dynamic surface exercise therapy; gross motor
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: 38 children with CP were randomly assigned to 2 groups. 1 group was interventional group and second group was control group. Both the groups were provided with therapy ( interventional group was provided with conventional therapy and intervention. control group was provided with conventional therapy only) and results were analyzed based on performance of both groups.
Who Masked: Outcomes Assessor
Masking Description: the outcome assessor was masked and had no idea about which participants were assigned to which group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dynamic surface exercise training group (Experimental): This group includes 19 subjects all of which are children with spastic diplegic cerebral palsy of GMFCS levels 3 and 4. This group received a set of exercises on various dynamic surfaces along with routine physical therapy. This group underwent a 60-minutes vigorous exercise program four days a week for two months
  Interventions: Other: Dynamic surface exercise training
- conventional physical therapy group (Active Comparator): This group includes 19 subjects all of which are children with spastic diplegic cerebral palsy of GMFCS levels 3 and 4. This group received only conventional physical therapy which is based upon principles of NDT. This group underwent a 60-minutes vigorous exercise program four days a week for two months.
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: Dynamic surface exercise training — Dynamic surface exercise training involves a set of exercises that are performed on various dynamic surfaces like gym ball and vestibular swing. All these exercise provide optimal arousal as they provide proprioceptive and vestibular stimulus. This group received a set of exercises on various dynamic surfaces.These exercises were implemented for 60 minutes for four days a week for two months.And it was observed how these exercises impacted gross motor function and trunk control of children with diplegic cerebral palsy of GMFCS level 3 and 4
  Arms: dynamic surface exercise training group
Other: conventional physical therapy — conventional physical therapy based on NDT involves a set of exercises that mostly include positioning exercises such as quadruped, side sitting, reaching sideways and overhead in sitting and catch and throw activities.
  Arms: conventional physical therapy group

SUMMARY:
The purpose of this study was to determine the effect of dynamic surface exercise treatment on trunk control and gross motor abilities in children with spastic diplegic cerebral palsy.

DETAILED DESCRIPTION:
A clinical trial was conducted to assess the impact dynamic surface exercise training on gross motor and trunk control of children with spastic diplegic cerebral palsy. The trial enrolled 38 children with spastic diplegic cerebral palsy of GMFCS levels 3 and 4. Children were randomly assigned to either the DSET or conventional physiotherapy training groups. Both groups underwent 60-minute vigorous exercise program four days a week for two months. The trunk control measurement scale was used to assess trunk control, while the GMFM-88 was used to assess gross motor function. Trunk control and gross motor function scores were obtained at the beginning, the fourth week, and the eighth week.

ELIGIBILITY:
Inclusion Criteria

* Diplegic children having Cerebral Palsy
* Children of age 5 - 12 years
* Children of GMFCS- E &R level III and IV
* Children who can follow verbal commands

Exclusion Criteria:

* Children with epileptic fits
* Children presenting with lower limb muscular contractures
* Children with scoliosis

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Gross motor function measure- 88 | change in baseline scores and 8th week scores
  The Gross Motor Function Measure (GMFM 88) is used to evaluate change that occurs over time in the gross motor function of children with cerebral palsy.
  It explores five areas of motor ability, which are known as dimensions:
  A) Lying and rolling B) Sitting C) Crawling and kneeling D) Standing E) Walking, running and jumping
trunk control measurement scale | change in baseline scores and 8th week scores
  The Trunk Control Measurement Scale is a clinical tool to measure trunk control in children with cerebral palsy. total score is 58 . low score means severely impaired trunk control and a high score shows better trunk control

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Hameed, DPT, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No